CLINICAL TRIAL: NCT05506280
Title: Association Between Prolactin Levels in Pregnant Women to- 2 Gether With Rates of Breastfeeding and the COVID-19 Virus. A 3 Randomised Trial
Brief Title: Association Between Prolactin Levels in Pregnant Women in COVID-19. Gether With Rates of Breastfeeding and the Covid-19 Virus
Status: Completed | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Other Study IDs: 16/08/22
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Breastfeeding; COVID-19 Infection
Keywords: Covid-19 infection; Pregnant women; Prolactin levels; Breastfeeeding
MeSH Terms: conditions — Breast Feeding; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: pregnant women infected by Covid-19
  Interventions: Procedure: blood prolactin levels

INTERVENTIONS:
Procedure: blood prolactin levels — The extraction technique was performed by venipuncture in 110 veins located in the antecubital area with a 21G butterfly nut with a Vacutainer Safety 111 Lok@ adapter, a 2.5x45cm latex venous compressor and a tube with separating gel 112 (yellow cap)

SUMMARY:
Background: Currently in the world, 41% of children under 6 months are exclusively breastfed. The Covid-19 pandemic has had a major impact on breastfeeding.; Methods: A statistical analysis of linear regression, prolactin analysis in the 3rd trimester of pregnancy and 15 days 15 after delivery was performed in women with Covid- 19 infection and healthy, finally the rates of 16 breastfeeding were evaluated. The sample was made up of 680 pregnant women from the Valladolid 17 Health Area, central region of Spain.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women under the coding of the clinical process of normal pregnancy or diagnosis of Covid-19 infection

Exclusion Criteria:

* No informed consent.
* No pregnant women.
* Older than 50 years old.
* Younger than 16 years old.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Study Population: pregnant women under the coding of the clinical process of normal pregnancy or diagnosis of Covid-19 infection
Sampling Method: Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Prolactin value | 15 days
  ng/ml. 0 mimimun, 100 maximum

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Humbwavali JB, Giugliani C, Silva ICMD, Duncan BB. Temporal trends in the nutritional status of women and children under five years of age in sub-Saharan African countries: ecological study. Sao Paulo Med J. 2018 Sep-Oct;136(5):454-463. doi: 10.1590/1516-3180.2017.0267261117. PMID 30570097
- [Result] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Result] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Result] Juan J, Gil MM, Rong Z, Zhang Y, Yang H, Poon LC. Effect of coronavirus disease 2019 (COVID-19) on maternal, perinatal and neonatal outcome: systematic review. Ultrasound Obstet Gynecol. 2020 Jul;56(1):15-27. doi: 10.1002/uog.22088. PMID 32430957
- [Result] Huntley BJF, Huntley ES, Di Mascio D, Chen T, Berghella V, Chauhan SP. Rates of Maternal and Perinatal Mortality and Vertical Transmission in Pregnancies Complicated by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Co-V-2) Infection: A Systematic Review. Obstet Gynecol. 2020 Aug;136(2):303-312. doi: 10.1097/AOG.0000000000004010. PMID 32516273
- [Result] Galang RR, Chang K, Strid P, Snead MC, Woodworth KR, House LD, Perez M, Barfield WD, Meaney-Delman D, Jamieson DJ, Shapiro-Mendoza CK, Ellington SR. Severe Coronavirus Infections in Pregnancy: A Systematic Review. Obstet Gynecol. 2020 Aug;136(2):262-272. doi: 10.1097/AOG.0000000000004011. PMID 32544146
- [Result] Rasmussen SA, Smulian JC, Lednicky JA, Wen TS, Jamieson DJ. Coronavirus Disease 2019 (COVID-19) and pregnancy: what obstetricians need to know. Am J Obstet Gynecol. 2020 May;222(5):415-426. doi: 10.1016/j.ajog.2020.02.017. Epub 2020 Feb 24. PMID 32105680